CLINICAL TRIAL: NCT04744584
Title: Optimizing Drug Management of Patients Suffering From Rare Disease Through Medication Reconciliation: Proof of Concept in Pulmonary Hypertension
Brief Title: Medication Reconciliation in Pulmonary Hypertension
Acronym: OPTICARE-HTP
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Agence Regionale de Sante d'Ile de France (Other Government)
Responsible Party: Sponsor
Other Study IDs: APHP201214; 2020-A02455-34 (Other: IDRCB)
Record Dates: First submitted 2021-01-15; First posted 2021-02-09 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Pulmonary Hypertension; Pulmonary Hypertension Chronic Thromboembolic; Pulmonary Arterial Hypertension
Keywords: pulmonary hypertension; medication reconciliation; medication errors; pharmacist; rare disease
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Arterial Hypertension; Rare Diseases | interventions — Medication Reconciliation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with medication reconciliation: Patient with medication reconciliation during 1st hospitalization
  Interventions: Other: Medication reconciliation
- Patients without medication reconciliation: Patient without medication reconciliation (MR) at 1st hospitalization but with retrospective MR at the next one (3 to 6 months after)
  Interventions: Other: Medication reconciliation

INTERVENTIONS:
Other: Medication reconciliation — MR will be performed directly upon entering the patient's hospital for a first PAH or HTP-Thrombo embolic assessment, just after inclusion. Information regarding the treatments taken by the patient at the time of admission will be retrieved. The entry medication assessment will then be compared with the first medical prescription in order to identify whether medications have been forgotten, prescribed at a different dosage or prescribed when not indicated, etc. All of these differences will be considered medication errors if the reason for the discrepancy is not entered in the patient medical file.
  Groups: Patients with medication reconciliation
Other: Medication reconciliation — After inclusion of the patient, the MR will be carried out retrospectively, that is to say that the information concerning the treatments taken by the patient at the time of the first assessment will be retrieved during the period of the first reassessment (therefore with a delay of 12 months depending on the deadline for the first assessment). All these discrepancies will be considered medication errors if the reason for the discrepancy was not entered in the patient's computerized medical record (IMR).
  Groups: Patients without medication reconciliation

SUMMARY:
Pulmonary hypertension (PH) is a life threatening condition. In PH, pulmonary arterial hypertension (PAH) and chronic thrombo-embolic chronic pulmonary hypertension (CTEPH) are two rare diseases requiring specific and complex drug management. In France ,a part of these treatments ,only available in hospital pharmacies, are generally unknown from community health care professionals despite the high risk of drug-interactions and side effects. Anticipating medication errors at the begging of the disease is therefore important, and could be done through medication reconciliation.

DETAILED DESCRIPTION:
Medication reconciliation (MR) will be done for patients hospitalized in the French referral center for PH for PAH or CTEPH. Detected medication errors will be tracked and fixed by the physician before the end of hospitalization. A synthesis of new/stopped and modified treatments will be given to the patient as well as his related healthcare professionals (community pharmacist and general practioner) to ensure the maintaining of the new therapeutic management and the understanding of drugs modification. To compare the potential decrease of medication errors promoted by MR, a retrospective MR will be also done for patients without MR at 1st hospitalization but at the next one (3 to 12 months after).

ELIGIBILITY:
Inclusion Criteria:

* Patient affiliated or entitled to a social security scheme
* At least 18 years old
* Patient with enlightened information of the study and not opposed with it.
* For patient without MR: patient hospitalized for the first re-evaluation of PAH or CTEPH within 12 months following the first assessment hospitalization (ie: first right heart catheterization at bicetre Hospital).
* For patient with MR: patient hospitalized for first assessment (first right heart catheterization at bicetre Hospital) of PAH or CTEPH

Exclusion Criteria:

* Patient suffering from another form of PH
* Patient under guardianship or curator
* Inability to give information to the patient either due to language barrier or to cognitive impairment
* Patient hosted in institution on discharge from hospital (follow-up care and long-term rehabilitation)
* Patient with a life expectancy of less than 1 year
* Patient on transplant list
* Patient refusal
* Length of stay < 48 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized in the French referal center to confirm PAH or CETPH diagnosis or coming back after diagnosis hospitalization
Sampling Method: Non-Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2021-02-16 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2024-06-15 (Actual)

PRIMARY OUTCOMES:
Proportion of patients having at least one medication error on discharge at the first hospitalization. | 12months
  This group will be compared to patients without prospective MR. For the latter group, MR is retrospective (3 to 6 months after discharge).

SECONDARY OUTCOMES:
Qualitative description of identified medication errors. | 12 months
  Omission, dosing errors, drug interactions, substitution of another active compound
Medication errors status | 12 Months
  corrected/not corrected
Identification of medication error severity | 12 months
  Cornish scale is the title of the scale which include 3 levels of gravity (from 1 to 3). The first one describes no relevant clinical impact and the third one describes a severe clinical impact.
Satisfaction of community healthcare practitioners with study tools | 12 months
  healthcare practitioners will be contacted by mail or phone
Therapeutic adherence | within 12 months after first hospitalization for the diagnosis of the disease
  Observance Girerd auto-questionnaire
Measure of Quality of life | within 12 months after first hospitalization for the diagnosis of the disease
  Short Form 36 Questionnaire
Improve vaccination coverage against influenza and pneumococcal disease | within 12 months after first hospitalization for the diagnosis of the disease
  inclusion vaccination coverage rate vs EOS(Enhanced Outreach Strategy) vaccination coverage rate
Emergency hospitalization | within 12 months after first hospitalization for the diagnosis of the disease
  Number of emergency hospitalizations between first assessment hospitalization (diagnosis) and first reassessment hospitalization
Estimate the time and resources spent on the conciliation process in the department | 12 months
  Time measurement of the conciliation process in the group with CM (in minutes)

CONTACTS AND LOCATIONS:
Overall Officials: Marie-camille CHAUMAIS, PharmaD, PHD, Principal Investigator — APHP
Locations (1):
- Hospital BICETRE, Le Kremlin-Bicêtre, France

IPD SHARING:
Plan to Share IPD: No
No sharing